CLINICAL TRIAL: NCT00542503
Title: Vascular Stiffness and Pulmonary Congestion
Brief Title: Using Magnetic Resonance Imaging to Predict People Who Are Likely to Develop Flash Pulmonary Edema (The PREDICT Study)
Acronym: PREDICT
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 478; R01HL076438-01A2 (NIH)
Record Dates: First submitted 2007-10-05; First posted 2007-10-11 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Heart Failure, Congestive
Keywords: Cardiac Outcomes; MRI; Cardiac Stress Testing
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Flash pulmonary edema is a sudden, abnormal build-up of fluid in the lungs. It is usually caused by heart failure and can be life threatening. The purpose of this study is to determine if a new form of magnetic resonance imaging (MRI) can identify abnormal blood flow to the lungs and predict increased risk of developing flash pulmonary edema among older adults.

DETAILED DESCRIPTION:
Pulmonary edema is a condition in which an abnormal build-up of fluid occurs in the lungs, which then leads to swelling. Symptoms include shortness of breath, breathing difficulty, and coughing. Flash pulmonary edema, which develops suddenly and can be life-threatening, is usually caused by heart failure. It occurs when the left ventricle of the heart is weakened and does not function properly, potentially impeding the flow of blood from the heart to the rest of the body. Blood pressure and fluid volume then increase, and excess blood accumulates in the blood vessels and tissues of the lungs. Flash pulmonary edema requires immediate treatment, including supplemental oxygen, mechanical ventilation, or medication. This study will determine if a new form of MRI testing can be used to identify probable abnormalities in blood flow to the lungs and predict increased risk of developing flash pulmonary edema among older adults.

This study will enroll people who are at risk of developing flash pulmonary edema. At a baseline study visit, participants will undergo a medical record review, a physical exam, blood collection, questions about cardiovascular health, and an MRI stress test. For the stress test, participants will first receive the medication dobutamine, which will increase their heart rate and reduce the blood supply to their heart. Participants will then be placed in an MRI machine and images of their heart will be taken. All participants will complete follow-up cardiovascular health questionnaires three times a year for 1 to 10 years, depending on when participants are enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be diagnosed with one of the following conditions:

  1. Diabetes with a fasting glucose level greater than or equal to 126 mg/dl and has been receiving treatment for more than 5 years
  2. High blood pressure with a history of a systolic blood pressure level greater than 140 mm Hg and a diastolic blood pressure level greater than 85 mm Hg while on medication
  3. Coronary artery disease

Exclusion Criteria:

* Prior heart attack encompassing greater than 5% of the left ventricular mass (total MB greater than 3 or Troponin I greater than 2)
* Heart attack, acute coronary syndrome (ACS), or angina within the 1 year prior to study entry
* Medical inability to use any cardiovascular magnetic resonance device (e.g., implanted electronic devices, intracranial metal, claustrophobia, closed angle glaucoma)
* Medically unable to receive dobutamine
* 3-vessel or left main coronary artery disease
* Moderate to severe valvular heart disease
* Left ventricular ejection fraction (LVEF) less than 25%
* History of pulmonary edema
* Serum creatinine level greater than 2.4 mg/dL or estimated glomerular filtration rate (eGFR) less than 30 mL/min
* Use of an investigational drug or device within the 30 days prior to study entry
* Diagnosed with any systemic disease, including cancer, with a reduced life expectancy of less than 12 months
* Chronic atrial fibrillation

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with diabetes, high blood pressure, or coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 579 (Actual)
Dates: Start 2007-06-01 (Actual); Primary Completion 2013-12-01 (Actual); Study Completion 2013-12-01 (Actual)

PRIMARY OUTCOMES:
Association between MRI stress measures of cardiovascular stiffness and cardiovascular events | Participants will be followed by phone for 5 years and up to 10 years pending renewal.

CONTACTS AND LOCATIONS:
Overall Officials: William G. Hundley, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Stacey RB, Vera T, Morgan TM, Jordan JH, Whitlock MC, Hall ME, Vasu S, Hamilton C, Kitzman DW, Hundley WG. Asymptomatic myocardial ischemia forecasts adverse events in cardiovascular magnetic resonance dobutamine stress testing of high-risk middle-aged and elderly individuals. J Cardiovasc Magn Reson. 2018 Nov 22;20(1):75. doi: 10.1186/s12968-018-0492-5. PMID 30463565
- [Derived] Vasu S, Little WC, Morgan TM, Stacey RB, Ntim WO, Hamilton C, Thohan V, Chiles C, Hundley WG. Mechanism of decreased sensitivity of dobutamine associated left ventricular wall motion analyses for appreciating inducible ischemia in older adults. J Cardiovasc Magn Reson. 2015 Apr 8;17(1):26. doi: 10.1186/s12968-015-0131-3. PMID 25885436
- [Derived] Vasu S, Morgan TM, Kitzman DW, Bertoni A, Stacey RB, Hamilton C, Chiles C, Thohan V, Hundley WG. Abnormal stress-related measures of arterial stiffness in middle-aged and elderly men and women with impaired fasting glucose at risk for a first episode of symptomatic heart failure. J Am Heart Assoc. 2015 Jan 14;4(1):e000991. doi: 10.1161/JAHA.114.000991. PMID 25589534
- [Derived] Jeevanantham V, Chughtai H, Little WC, Morgan T, Kitzman DW, Hamilton CA, Hundley WG. Aging reduces left atrial performance during adrenergic stress in middle aged and older patients. Cardiol J. 2012;19(1):45-52. doi: 10.5603/cj.2012.0008. PMID 22298167
- [Derived] Chughtai HL, Morgan TM, Rocco M, Stacey B, Brinkley TE, Ding J, Nicklas B, Hamilton C, Hundley WG. Renal sinus fat and poor blood pressure control in middle-aged and elderly individuals at risk for cardiovascular events. Hypertension. 2010 Nov;56(5):901-6. doi: 10.1161/HYPERTENSIONAHA.110.157370. Epub 2010 Sep 13. PMID 20837881